CLINICAL TRIAL: NCT03268811
Title: A Prospective, Open-label, Long-term Safety and Efficacy Study of Teduglutide in Japanese Pediatric Subjects With Short Bowel Syndrome Who Completed SHP633-302
Brief Title: A Study in Japanese Children With Short Bowel Syndrome Who Completed SHP633-302
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHP633-305; 2021-005404-36 (EudraCT Number)
Record Dates: First submitted 2017-08-10; First posted 2017-08-31 (Actual); Results first posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-04

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Teduglutide (Experimental): Participants will receive teduglutide 0.05 milligram per kilogram (mg/kg) subcutaneous (SC) injection once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm for 24-week intervals. If a participant deteriorates during a follow-up period, the participant may be evaluated immediately for additional teduglutide treatment (24-week interval) until teduglutide is commercially available for each participant, the participant's participation in this study is discontinued, or the study is discontinued.
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Teduglutide 0.05 mg/kg SC injection will be administered once daily into 1 of the 4 quadrants of the abdomen or either thigh or arm.

SUMMARY:
The purpose of this clinical study is to evaluate the long-term safety and tolerability of teduglutide treatment in Japanese pediatric participants with short bowel syndrome (SBS) who completed Study SHP633-302 (NCT02980666).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by a parent or guardian prior to any study-related procedures.
* When applicable, informed assent (as deemed appropriate by the Institutional Review Board [IRB]) by the participant prior to any study-related procedures.
* Participant completed Study SHP633-302 (NCT02980666).
* Participant (and/or parent/guardian) understands and is willing and able to fully adhere to study requirements as defined in this protocol.

Exclusion Criteria:

There are no exclusion criteria for this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (6):
- Japan (6):
  - Akita University Hospital, Akita, Akita
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Tsukuba University Hospital, Tsukuba, Ibaraki
  - Kagoshima University Hospital, Kagoshima, Kagoshima-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - Showa University Hospital, Shinagawa-ku, Tokyo-To

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …).

REFERENCES:
- [Derived] Chiba M, Masumoto K, Kaji T, Matsuura T, Morii M, Fagbemi A, Hill S, Pakarinen MP, Protheroe S, Urs A, Chen ST, Sakui S, Udagawa E, Wada M. Efficacy and Safety of Teduglutide in Infants and Children With Short Bowel Syndrome Dependent on Parenteral Support. J Pediatr Gastroenterol Nutr. 2023 Sep 1;77(3):339-346. doi: 10.1097/MPG.0000000000003867. Epub 2023 Jun 26. PMID 37364133
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fd94db2bf003ab470dd

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in Japan from 23 August 2017 (first participant first visit) and 02 November 2021 (last participant last visit).
Pre-assignment Details: A total of 9 Japanese pediatric participants who completed Study SHP633-302 (NCT02980666) were enrolled into the extension study based on age of participants i.e., 7 children (aged 1 through 15 years of age) and 2 infants (aged 4 months through < 12 months of corrected gestational age).
Groups:
- Total Children (Aged: 1 to 15 Years): Participants aged from 1 through 15 years who participated in the core study (SHP633-302 [NCT02980666]) were enrolled into this extension study and received teduglutide 0.05 milligram per kilogram (mg/kg) subcutaneous (SC) injection once daily for 24 weeks in each treatment cycle depending on the disease course.
- Infants (Corrected Gestational Age: 4 to < 12 Months): Participants (Infants) from 4 through < 12 months of corrected gestational age who participated in the core study (SHP633-302 [NCT02980666]) were enrolled into this extension study and received teduglutide 0.05 mg/kg SC injection once daily for 24 weeks in each treatment cycle depending on the disease course.
Period: Overall Study
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Started | 7 | 2
Completed | 7 | 1
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]).
Groups:
- Total Children (Aged: 1 to 15 Years): Participants aged from 1 through 15 years who participated in the core study (SHP633-302 [NCT02980666]) were enrolled into this extension study and received teduglutide 0.05 mg/kg SC injection once daily for 24 weeks in each treatment cycle depending on the disease course.
- Total: Total of all reporting groups
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months) | Total
Number analyzed (Participants) | 7 | 2 | 9
Age, Customized [Count of Participants; unit: Participants]
  Aged: 1 to 15 Years | 7 | 0 | 7
  Aged: 4 to < 12 Months | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as any AEs whose onset occurred, severity worsened or intensity increased after receiving the investigational product (IP) in the core study (SHP633-302 [NCT02980666]) or this extension study. Number of participants with TEAEs were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: From Baseline up to follow-up (up to 50 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 2
Participants | 7 | 2

2. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital sign assessments included pulse rate, blood pressure (systolic and diastolic blood pressure) and body temperature. Number of participants with clinically significant abnormalities in vital signs which were deemed clinically significant by the investigator were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: From Baseline up to follow-up (up to 50 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 2
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Clinical laboratory parameters included biochemistry, hematology and urinalysis. Number of participants with clinically significant abnormalities in laboratory parameters which were deemed clinically significant by the investigator were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: From Baseline up to follow-up (up to 50 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Infants (Corrected Gestational Age: 4 to < 12 Months): Participants (Infants) from 4 through < 12 months of corrected gestational age who participated in the core study (SHP633-302 [NCT02980666]) were enrolled into this extension study and received teduglutide 0.05 mg/kg SC injection once daily for 24 weeks in each treatment cycle (Cycles 1 to 9 [Each cycle=28 weeks]) depending on the disease course.
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 7 | 2
Participants
  Biochemistry | 5 | 1
  Hematology | 1 | 0
  Urinalysis. | 0 | 0

4. Primary Outcome: Percent Change From Baseline in Average Total Urine Output at End of Treatment (EOT) of Last Cycle During Teduglutide Treatment
Description: Average total urine output was recorded over a 48-hour period of parental support (PS) stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The Average daily urine output milliliter per kilogram per day (mL/kg/day) was calculated as: (Total urine output over 48 hours / 2) / body weight (kilogram [kg]) where total urine output was calculated as the sum of the urine output in milliliter (mL) and the urine-only diaper weights in gram (g) (1g = 1mL) for the participant collected on the output diary form of electronic case report from (eCRF). Percent change from baseline in average total urine output at EOT of last cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Percent change | -37.228 (42.9396) | 146.881 (295.8061)

5. Primary Outcome: Percent Change From Baseline in Average Number of Stools Per Day at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized by the average number of stools per day. The average number of stools per day was calculated as (sum of the daily data in a 48-hour period/2). Percent change from baseline in average number of stools per day at EOT of last cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Percent change | 24.37 (63.623) | 50.00 (0.000)

6. Primary Outcome: Percent Change From Baseline in Average Stool/Mixed Stool Diaper Weight at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized by the average stool/mixed stool diaper weight (gram per kilogram per day [g/kg/day]). The body weight was used to calculate the daily stool/mixed stool diaper weight (g/kg/day). Percent change from baseline in average stool/mixed stool diaper weight at EOT of last cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 1 | 2
Percent change | -12.678 (NA) — Standard deviation could not be calculated because single participant was analyzed. | 206.017 (332.4580)

7. Primary Outcome: Percent Change From Baseline in Average Total Ostomy Output at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The body weight was used to calculate the average total ostomy output per day (mL/kg/day) using a formula analogous to that used to calculate the average daily urine output. Percent change from baseline in average total ostomy output at EOT of last cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here, "0" in Overall number of participants analyzed signifies that no participant was evaluable at specified time point for the specified group.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 2
Percent change |  | 3.143 (145.8659)

8. Primary Outcome: Percent Change From Baseline in Average Bristol Stool Form Score at EOT of Last Cycle During Teduglutide Treatment
Description: Fecal output was recorded over a 48-hour period of PS stability before every scheduled site visit and within 1 week of implementing any PS adjustment. The average daily fecal output was summarized the average typical stool form score using Bristol Stool Form Scale. The average typical stool form score was calculated as (sum of the daily data in a 48-hour period / 2). Typical Stool Form based on Bristol Stool Form Scale: 1 - Separate hard lumps, hard to pass, 2 - Sausage-shaped, but lumpy, 3 - Like a sausage but with cracks on the surface, 4- Like a sausage or snake, smooth and soft, 5- Soft blobs with clear-cut edges, 6- Fluffy pieces with ragged edges, a mushy stool, 7- Watery, no solid pieces. Entirely liquid. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]). A negative change from baseline indicates improvement.
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Percent change | -7.51 (16.758) | 0.00 (0.000)

9. Primary Outcome: Number of Participants With Anti-drug Antibodies (ADAs) (Including Neutralizing Antibodies) at EOT of Last Cycle During Teduglutide Treatment
Description: Number of participants with ADAs (including NAbs) to teduglutide were used to summarize the presence of antibodies. The participants who tested positive only for ADAs (including NAbs) were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "overall number of participants analyzed" refer to the participants evaluable for this outcome measure and "number analyzed" refer to participants evaluable for this outcome at given categories. "0" in number analyzed signifies that no participant was evaluable for specified category for the specified group.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Participants
  Positive ADA at EOT of the Last Cycle | 5 | 0
  Positive NAbs at EOT of the Last Cycle: number analyzed (Participants) | 5 | 0
  Positive NAbs at EOT of the Last Cycle | 4 |

10. Primary Outcome: Number of Participants With Clinically Significant Changes in Gastrointestinal (GI) Specific Testing
Description: GI specific testing included colonoscopy or sigmoidoscopy, abdominal ultrasound, fecal occult blood testing, upper GI series with small bowel follow-through (UGI/SBFT). Number of participants with clinically significant changes findings in gastrointestinal specific testing were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Participants | 0 | 0

11. Primary Outcome: Change From Baseline in Body Weight For Age Z-Score at EOT of Last Cycle During Teduglutide Treatment
Description: Body weight was measured using Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in body weight for age Z-Score at EOT of last cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of last cycle (up to Month 45) (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Z-score | 0.229 (0.5636) | 3.982 (3.6363)

12. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 1 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-Score at EOT of cycle 1 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 1 (up to 24 Weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Z-score | 0.002 (0.6049) | 1.376 (0.3363)

13. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 2 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 2 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 2 (up to 48 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 1
Z-score | 0.152 (0.5181) | 3.114 (NA) — Standard deviation could not be calculated because single participant was analyzed.

14. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 3 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 3 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 3 (up to 72 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 1
Z-score | 0.098 (0.3467) | 3.554 (NA) — Standard deviation could not be calculated because single participant was analyzed.

15. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 4 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 4 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 4 (up to 96 weeks)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Z-Score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 5 | 1
Z-Score | 0.126 (0.2622) | 3.542 (NA) — Standard deviation could not be calculated because single participant was analyzed.

16. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 5 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 5 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 5 (up to 120 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here,"0" in Overall number of participants analyzed signifies that no participant was evaluable at specified time point for the specified group.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 3 | 0
Z-score | 0.342 (0.1012) |

17. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 6 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 6 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 6 (up to 144 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 2 | 0
Z-score | 0.276 (0.2593) |

18. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 7 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 7 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 7 (up to 168 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 1 | 0
Z-score | 0.570 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

19. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 8 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 8 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 8 (up to 192 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 1 | 0
Z-score | 0.851 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

20. Primary Outcome: Change From Baseline in Height For Age Z-Score at EOT of Cycle 9 During Teduglutide Treatment
Description: Height was measured using Age Z-Score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in height for age Z-score at EOT of Cycle 9 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 9 (up to 196 weeks)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 1 | 0
Z-score | 0.477 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

21. Primary Outcome: Change From Baseline in Head Circumference for Age Z-score at EOT of Cycle 1 During Teduglutide Treatment
Description: Head circumference was measured using Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in head circumference for Age Z-score at EOT of Cycle 1 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 1 (up to 24 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here, head circumference was collected only for participants with less than (<) 12 months of age.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 2
Z-score |  | 2.400 (0.6472)

22. Primary Outcome: Change From Baseline in Head Circumference for Age Z-score at EOT of Cycle 2 During Teduglutide Treatment
Description: Head circumference was measured using Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in head circumference for Age Z-score at EOT of Cycle 2 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 2 (up to 48 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here, head circumference was collected only for participants with < 12 months of age.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 1
Z-score |  | 1.431 (NA) — Standard deviation could not be calculated because single participant was analyzed.

23. Primary Outcome: Change From Baseline in Head Circumference for Age Z-score at EOT of Cycle 3 During Teduglutide Treatment
Description: Head circumference was measured using Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in head circumference for Age Z-score at EOT of Cycle 3 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 3 (up to 72 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 1
Z-score |  | 2.080 (NA) — Standard deviation could not be calculated because single participant was analyzed.

24. Primary Outcome: Change From Baseline in Head Circumference for Age Z-score at EOT of Cycle 4 During Teduglutide Treatment
Description: Head circumference was measured using Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in head circumference for Age Z-score at EOT of Cycle 4 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 4 (up to 76 weeks)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 0 | 1
Z-score |  | 2.055 (NA) — Standard deviation could not be calculated because single participant was analyzed.

25. Primary Outcome: Change From Baseline in Body Mass Index (BMI) for Age Z-score at EOT of Cycle 1 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 1 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 1 (up to 24 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here, BMI was calculated only for participants greater than or equal to (>=) 2 years of age.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 0
Z-score | 0.090 (0.6642) |

26. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 2 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 2 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 2 (up to 48 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, "Overall number of participants analyzed" signifies those participants who were evaluable for this outcome measure. Here, BMI was calculated only for participants >= 2 years of age.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 0
Z-score | 0.489 (0.8474) |

27. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 3 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 3 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 3 (up to 72 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 0
Z-score | 0.409 (1.1688) |

28. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 4 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 4 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 4 (up to 96 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 5 | 0
Z-score | 0.118 (0.8827) |

29. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 5 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 5 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 5 (up to 120 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 3 | 0
Z-score | 0.070 (0.9770) |

30. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 6 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 6 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 6 (up to 144 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 2 | 0
Z-score | 0.925 (0.2556) |

31. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 7 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 7 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 7 (up to 168 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 1 | 0
Z-score | 0.839 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

32. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 8 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 8 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 8 (up to 192 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 1 | 0
Z-score | 0.015 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

33. Primary Outcome: Change From Baseline in BMI for Age Z-score at EOT of Cycle 9 During Teduglutide Treatment
Description: BMI Z-score was calculated by using the height and weight Age Z-score. A Z-score was the deviation of the value for an individual from the mean value of the reference population divided by the standard deviation for the reference population. Centers for Disease Control and Prevention (age >= 2 years old) and World Health Organization (age < 2 years old) Z-score calculation charts were used for calculation. A negative Z-score indicates values lower than the mean while a positive Z-score indicates values higher than the mean. Change from baseline in BMI for Age Z-score at EOT of Cycle 9 during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of Cycle 9 (up to 196 weeks)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 1 | 0
Z-score | 0.480 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

34. Secondary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Reduction From Baseline in Participants Diary Parenteral Support (PS) Volume at EOT of Each Cycle During Teduglutide Treatment
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume during the treatment period. Percent reduction in weight-normalized diary PS values from baseline was calculated using the formula: % reduction in PS value at the visit = ([average daily value at the scheduled visit - average daily value at baseline of the core study (SHP633-302 [NCT02980666]) / average daily value at baseline of the core study (SHP633-302 [NCT02980666])) *100. Number of participants who achieved at least 20% reduction from baseline in participants diary PS volume at EOT of each cycle during teduglutide treatment were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: The safety population included all enrolled participants in the study and who received at least one dose of teduglutide (in study SHP633-302 [NCT02980666] or SHP633-305 [NCT03268811]). Here, overall number of participants analyzed signifies to the participants evaluable for this outcome measure and "number analyzed" signifies to participants evaluable for this outcome at given timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Participants
  At least 20% Reduction: At EOT of Cycle 1 | 4 | 1
  At least 20% Reduction: At EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  At least 20% Reduction: At EOT of Cycle 2 | 4 | 1
  At least 20% Reduction: At EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  At least 20% Reduction: At EOT of Cycle 3 | 6 | 1
  At least 20% Reduction: At EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  At least 20% Reduction: At EOT of Cycle 4 | 5 | 1
  At least 20% Reduction: At EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  At least 20% Reduction: At EOT of Cycle 5 | 3 |
  At least 20% Reduction: At EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  At least 20% Reduction: At EOT of Cycle 6 | 2 |
  At least 20% Reduction: At EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  At least 20% Reduction: At EOT of Cycle 7 | 1 |
  At least 20% Reduction: At EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  At least 20% Reduction: At EOT of Cycle 8 | 1 |
  At least 20% Reduction: At EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  At least 20% Reduction: At EOT of Cycle 9 | 1 |

35. Secondary Outcome: Number of Participants Who Achieved At Least 20 Percent (%) Reduction From Baseline in Investigator Prescribed PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume during the treatment period. Percent reduction in weight-normalized prescribed PS values from baseline was calculated using the formula: % reduction in PS value at the visit =([average daily value at the scheduled visit - average daily value at baseline of the core study (SHP633-302 [NCT02980666]) / average daily value at baseline of the core study (SHP633-302 [NCT02980666])) *100. Number of participants who achieved at least 20% reduction from baseline in Investigator prescribed PS volume at EOT of each cycle during teduglutide treatment were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Participants
  At least 20% Reduction: At EOT of Cycle 1 | 5 | 1
  At least 20% Reduction: At EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  At least 20% Reduction: At EOT of Cycle 2 | 5 | 1
  At least 20% Reduction: At EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  At least 20% Reduction: At EOT of Cycle 3 | 6 | 1
  At least 20% Reduction: At EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  At least 20% Reduction: At EOT of Cycle 4 | 5 | 1
  At least 20% Reduction: At EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  At least 20% Reduction: At EOT of Cycle 5 | 3 |
  At least 20% Reduction: At EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  At least 20% Reduction: At EOT of Cycle 6 | 2 |
  At least 20% Reduction: At EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  At least 20% Reduction: At EOT of Cycle 7 | 1 |
  At least 20% Reduction: At EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  At least 20% Reduction: At EOT of Cycle 8 | 1 |
  At least 20% Reduction: At EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  At least 20% Reduction: At EOT of Cycle 9 | 1 |

36. Secondary Outcome: Change From Baseline in Participant Diary PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume during the treatment period. Change from baseline in participants diary PS volume at EOT of each cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
mL/kg/day
  Change at EOT of Cycle 1 | -21.5 (11.83) | -31.9 (16.24)
  Change at EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 2 | -25.5 (14.38) | -54.2 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 3 | -32.1 (18.19) | -62.8 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  Change at EOT of Cycle 4 | -37.2 (24.10) | -95.8 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  Change at EOT of Cycle 5 | -54.8 (26.58) |
  Change at EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  Change at EOT of Cycle 6 | -63.8 (31.57) |
  Change at EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 7 | -93.8 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 8 | -80.3 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 9 | -79.1 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

37. Secondary Outcome: Percent Change From Baseline in Participant Diary PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume during the treatment period. Percent change from baseline in participants diary PS volume at EOT of each cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Percent change
  Percent change at EOT of Cycle 1 | -39.6 (34.86) | -32.5 (18.10)
  Percent change at EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  Percent change at EOT of Cycle 2 | -44.3 (33.11) | -56.6 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  Percent change at EOT of Cycle 3 | -52.8 (28.54) | -65.6 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  Percent change at EOT of Cycle 4 | -62.9 (26.18) | -100.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  Percent change at EOT of Cycle 5 | -73.9 (5.30) |
  Percent change at EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  Percent change at EOT of Cycle 6 | -75.7 (0.54) |
  Percent change at EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  Percent change at EOT of Cycle 7 | -82.9 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Percent change at EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  Percent change at EOT of Cycle 8 | -70.9 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Percent change at EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  Percent change at EOT of Cycle 9 | -69.8 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

38. Secondary Outcome: Change From Baseline in Investigator Prescribed PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume during the treatment period. Change from baseline in investigator prescribed PS volume at EOT of each cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: mL/kg/day
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
mL/kg/day
  Change at EOT of Cycle 1 | -20.9 (11.06) | -31.3 (26.77)
  Change at EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 2 | -28.0 (13.51) | -60.6 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 3 | -34.8 (21.13) | -67.5 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  Change at EOT of Cycle 4 | -36.3 (23.52) | -98.7 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  Change at EOT of Cycle 5 | -53.3 (26.24) |
  Change at EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  Change at EOT of Cycle 6 | -63.6 (32.10) |
  Change at EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 7 | -91.8 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 8 | -77.3 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 9 | -77.9 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

39. Secondary Outcome: Percent Change From Baseline in Investigator Prescribed PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: PS (parenteral nutrition or intravenous fluids) was considered for managing nutritional support in terms of volume during the treatment period. Percent change from baseline in investigator prescribed PS volume at EOT of each cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Percent change
  Percent change at EOT of Cycle 1 | -38.8 (35.19) | -32.1 (26.51)
  Percent change at EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  Percent change at EOT of Cycle 2 | -46.9 (30.42) | -61.4 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  Percent change at EOT of Cycle 3 | -55.4 (27.78) | -68.3 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  Percent change at EOT of Cycle 4 | -62.5 (26.45) | -100.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Percent change at EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  Percent change at EOT of Cycle 5 | -73.3 (5.51) |
  Percent change at EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  Percent change at EOT of Cycle 6 | -76.3 (2.41) |
  Percent change at EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  Percent change at EOT of Cycle 7 | -83.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Percent change at EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  Percent change at EOT of Cycle 8 | -69.9 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Percent change at EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  Percent change at EOT of Cycle 9 | -70.5 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

40. Secondary Outcome: Number of Participants Who Achieved Enteral Autonomy PS Volume at EOT of Each Cycle During Teduglutide Treatment
Description: Enteral autonomy (completely weaned off PS) was defined as the first visit where there is no use of PS for the 7 days prior to the visit and there is no prescribed PS at that visit, and the participants remains off PS for the remainder of the treatment period of that cycle. Number of participants who achieved enteral autonomy off PS volume at EOT of each cycle during teduglutide treatment were reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Participants
  At EOT of Cycle 1 | 1 | 0
  At EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  At EOT of Cycle 2 | 1 | 0
  At EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  At EOT of Cycle 3 | 1 | 0
  At EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  At EOT of Cycle 4 | 1 | 1
  At EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  At EOT of Cycle 5 | 0 |
  At EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  At EOT of Cycle 6 | 0 |
  At EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  At EOT of Cycle 7 | 0 |
  At EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  At EOT of Cycle 8 | 0 |
  At EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  At EOT of Cycle 9 | 0 |

41. Secondary Outcome: Change From Baseline in Days Per Week of Diary PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Days per week of diary PS was calculated as: Days per week of actual PS = (number of days with non-zero values for PS volume within the 7 days prior to the visit / number of days for which any PS intake data was recorded within the 7 days prior to the visit) * 7. Change from baseline in days per week of diary PS usage at EOT of each cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Days/week
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Days/week
  Change at EOT of Cycle 1 | -1.2 (2.86) | 0.0 (0.00)
  Change at EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 2 | -1.2 (2.86) | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 3 | -1.2 (2.86) | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  Change at EOT of Cycle 4 | -1.4 (3.13) | -7.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  Change at EOT of Cycle 5 | 0.0 (0.00) |
  Change at EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  Change at EOT of Cycle 6 | 0.0 (0.00) |
  Change at EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 7 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 8 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 9 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

42. Secondary Outcome: Change From Baseline in Days Per Week of Prescribed PS Usage at EOT of Each Cycle During Teduglutide Treatment
Description: Change from baseline in days per week of prescribed PS usage at EOT of each cycle during teduglutide treatment was reported. Days per week of diary PS was calculated as: Days per week of actual PS = (number of days with non-zero values for PS volume within the 7 days prior to the visit / number of days for which any PS intake data was recorded within the 7 days prior to the visit) * 7. Change from baseline in days Per week of prescribed PS usage at EOT of each cycle during teduglutide treatment was reported. Baseline refers to the baseline value of the core study (SHP633-302 [NCT02980666]).
Time Frame: Baseline, EOT of each cycle 1, 2, 3, 4, 5, 6, 7, 8 and 9 (Each Cycle 1 to 8 = 24 weeks, and Cycle 9 = 4 weeks)
Population: as for outcome 34
Measure: Mean (Standard Deviation); unit: Days/week
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
Number analyzed (Participants) | 6 | 2
Days/week
  Change at EOT of Cycle 1 | -1.2 (2.86) | 0.0 (0.00)
  Change at EOT of Cycle 2: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 2 | -1.2 (2.86) | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 3: number analyzed (Participants) | 6 | 1
  Change at EOT of Cycle 3 | -16.7 (40.82) | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 4: number analyzed (Participants) | 5 | 1
  Change at EOT of Cycle 4 | -20.0 (44.72) | -100.0 (NA) — Standard deviation could not be calculated because single participant was analyzed.
  Change at EOT of Cycle 5: number analyzed (Participants) | 3 | 0
  Change at EOT of Cycle 5 | 0.0 (0.00) |
  Change at EOT of Cycle 6: number analyzed (Participants) | 2 | 0
  Change at EOT of Cycle 6 | 0.0 (0.00) |
  Change at EOT of Cycle 7: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 7 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 8: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 8 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. |
  Change at EOT of Cycle 9: number analyzed (Participants) | 1 | 0
  Change at EOT of Cycle 9 | 0.0 (NA) — Standard deviation could not be calculated because single participant was analyzed. |

ADVERSE EVENTS:
Time Frame: From Baseline up to follow-up (up to 50 months)
Arm/Group | Total Children (Aged: 1 to 15 Years) | Infants (Corrected Gestational Age: 4 to < 12 Months)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/2
Serious Adverse Events (participants affected / at risk) | 7/7 | 2/2
Other Adverse Events (participants affected / at risk) | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Children (Aged: 1 to 15 Years) (N=7) | Infants (Corrected Gestational Age: 4 to < 12 Months) (N=2)
Colonic haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 4 (6) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Medical device site infection (Infections and infestations) | 1 (3) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 3 (8) | 1 (2)
Device damage (Product Issues) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Central venous catheter removal (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Children (Aged: 1 to 15 Years) (N=7) | Infants (Corrected Gestational Age: 4 to < 12 Months) (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (2) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
Strabismus (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (5) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Food allergy (Immune system disorders) | 1 (4) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Adenoviral conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (3)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Medical device site infection (Infections and infestations) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 4 (25) | 1 (5)
Auricular haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Epiphyseal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (6) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypozincaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (5) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Device damage (Product Issues) | 1 (1) | 0 (0)
Head banging (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT03268811/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT03268811/SAP_001.pdf